CLINICAL TRIAL: NCT03801265
Title: A Prospective, Randomized, Double-blinded, Active-comparator, Non-inferiority Study to Observe Relative Efficacy of Ultrasound-guided Transmuscular Quadratus Lumborum Block Versus Class Lumbar Plexus Block in Managing Post-operative Pain Following Total Hip Replacement Surgery
Brief Title: Lumbar Plexus vs Quadratus Lumborum Block in Post-operative Pain Following Total Hip Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sharad Khetarpal (Other)
Responsible Party: Sponsor-Investigator, Sharad Khetarpal, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO18120275
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Hip Osteoarthritis
Keywords: lumbar plexus block; quadratus lumborum block; total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Lumbar plexus block vs Quadratus lumborum type 3 block
Who Masked: Participant, Outcomes Assessor
Masking Description: The person who perform the block will be unblinded. The participants and the outcomes assessor will be blinded to the treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lumbar Plexus block (Active Comparator): 0.5% ropivacaine 100 mg (20 ml) will be injected
  Interventions: Procedure: Lumbar plexus block; Drug: Ropivacaine injection
- Quadratus Lumborum type 3 block (Experimental): 0.5% ropivacaine 100 mg (20 ml) will be injected
  Interventions: Procedure: Quadratus lumborum type 3 block; Drug: Ropivacaine injection

INTERVENTIONS:
Procedure: Lumbar plexus block — Patient will be positioned in lateral decubitus position with side to be blocked facing upwards. Midline will be identified by palpating the spinous process. Intercristal line will be drawn connecting iliac crests. The point of needle insertion will be 4 cm lateral to the intersection of both lines. The transverse process will first contact with a finder needle. Subsequently an 18 gauge 10 cm insulated needle will be used and advanced until it contacted the transverse process. Needle will then be redirected cephalad or caudad and advanced 2 cm, until the quadriceps femoris twitch is obtained. Local anesthetic will then be injected after confirming a motor response between 0.3-0.5 milli amperes.
  Arms: Lumbar Plexus block
Procedure: Quadratus lumborum type 3 block — Patient will be placed in a lateral position with the side to be blocked facing up. A low frequency transducer will be used to identify three layers of abdominal musculature, probe will be then moved posteriorly till the transverse abdominus aponeurosis is visualized, the QL muscle is then identified by tracing the aponeurosis posteriorly. The transducer is then moved more posteriorly to visualize the shadow of transverse process and the origin of QL muscle. Psoas muscle is then identified lying anterior to the QL muscle. A 22 gauge 8 cm is inserted in plane posterior to the probe and advanced intramuscularly through the QL to interfacial plane between QL and psoas major and local anesthetic is deposited.
  Arms: Quadratus Lumborum type 3 block
Drug: Ropivacaine injection — 0.5% ropivacaine 20 ml (100 mg) will be injected for both groups.

SUMMARY:
The Lumbar Plexus (LP) block is currently used as the standard-of-care regional anesthesia technique to provide postoperative pain management after primary hip replacement surgery at UPMC Shadyside Hospital. However, the LP technique is complex and can be associated with potentially serious side effects, including nerve injury, major bleeding, retroperitoneal hematoma, and intrathecal injection of local anesthetic. In rare instances the LP block can also lead to motor blockade, interfering with early ambulation. There are several case reports of Quadratus Lumborum inter-fascial block (QL3) giving equally adequate pain relief after total hip replacement surgery, and this QL3 block is performed routinely at this institution. The benefits to inter-fascial administration of local anesthetic include the avoidance of theoretical nerve injury, bleeding and intrathecal anesthetic administration associated with the direct interaction between the nerve and the nerve block needle. The purpose of this study is to show that QL3 block is non-inferior to the standard-of-care lumbar plexus block and should be used more regularly in hip replacement surgery. The study will be conducted as a prospective, randomized (1:1), double-blind, non-inferiority, active-comparator trial. The investigators plan to enroll 40 subjects, 20 in each treatment group. This study will prospectively investigate the efficacy of QL3 versus Classic LP block for post-operative pain management in subjects undergoing primary, unilateral hip replacement surgery and prospectively compare QL3 versus Classic LP block in time to mobilization and physical therapy response. Primary outcome measures include pain at rest and with movement at 6, 12 and 24 hours after surgery. Secondary outcomes will be time for first request for pain medication, total pain medications (narcotics and non-narcotic analgesics) given in 24 hours and the time of participant's ability to walk 100 feet as recorded by a physical therapist.

DETAILED DESCRIPTION:
Eligible patients will be approached for the study by the PI or Sub-I in the pre-operative area on their day of surgery. The anesthesiology investigator will speak with the patient about the study behind a closed drape and the patient will have adequate time to consider the consent and ask questions regarding risk factors associated with each type of block. Once consented, the patient will be randomized by computer generated random number to one of the two treatment groups. Once assigned the treatment allocation, only the clinician administering the block will be unblinded to the randomization outcome. If randomized to the LP block, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach: Patient will be positioned in lateral decubitus position with side to be blocked facing upwards. Midline will be identified by palpating the spinous process. Intercristal line will be drawn connecting iliac crests. The point of needle insertion will be 4 cm lateral to the intersection of both lines. The transverse process will first contact with a finder needle. Subsequently an 18 gauge 10 cm insulated needle will be used and advanced until it contacted the transverse process. Needle will then be redirected cephalad or caudad and advanced 1 cm, until the quadriceps femoris twitch is obtained. Local anesthetic will then be injected after confirming a motor response between 0.3-0.5 milli amperes.If randomized to the QL3 block, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach:Patient will be placed in a lateral position with the side to be blocked facing up. A low frequency transducer will be used to identify three layers of abdominal musculature, probe will be then moved posteriorly till the transverse abdominus aponeurosis is visualized, the QL muscle is then identified by tracing the aponeurosis posteriorly. The transducer is then moved more posteriorly to visualize the shadow of transverse process and the origin of QL muscle. Psoas muscle is then identified lying anterior to the QL muscle. A 22 gauge 8 cm is inserted in plane posterior to the probe and advanced intramuscularly through the QL to interfacial plane between QL and psoas major and local anesthetic is deposited. For both treatment groups, the local anesthetic used will be 100 mg 0.5% ropivacaine. After surgery, the patient will be followed by the blinded research team for incidence of adverse events, as well as the collection of the primary outcome measures. These include pain at rest and with movement at 6, 12 and 24 hours after surgery, time for first request for pain medication, total pain medications (narcotics and non-narcotic analgesics) given in 24 hours and the time of participant's ability to walk 100 feet as recorded by physical therapist. This information will be captured from the patient's electronic medical record.

Minor changes were made to the outcome measures after the original approval of this submission. This was only to clarify the specific measures from the more general descriptions in the original.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-90 years old
2. Primary unilateral total hip arthroplasty
3. BMI 20 - 36
4. Male and Female
5. All races

Exclusion Criteria:

1. Patient refusal
2. ASA class > or = 4
3. Pregnancy
4. Any condition precluding patient going home with in 24 hours of surgery
5. Non-English speaking or inability to participate in the study
6. Patients with coagulopathy or on therapeutic anticoagulation
7. Chronic Steroid Use
8. Narcotic Addiction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharad Khetarpal, MD, Principal Investigator — Department of Anesthesiology, University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian-Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilfeld BM, Ball ST, Gearen PF, Le LT, Mariano ER, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Meyer RS. Ambulatory continuous posterior lumbar plexus nerve blocks after hip arthroplasty: a dual-center, randomized, triple-masked, placebo-controlled trial. Anesthesiology. 2008 Sep;109(3):491-501. doi: 10.1097/ALN.0b013e318182a4a3. PMID 18719448
- [Background] Weller RS, Gerancher JC, Crews JC, Wade KL. Extensive retroperitoneal hematoma without neurologic deficit in two patients who underwent lumbar plexus block and were later anticoagulated. Anesthesiology. 2003 Feb;98(2):581-5. doi: 10.1097/00000542-200302000-00044. No abstract available. PMID 12552223
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Hockett MM, Hembrador S, Lee A. Continuous Quadratus Lumborum Block for Postoperative Pain in Total Hip Arthroplasty: A Case Report. A A Case Rep. 2016 Sep 15;7(6):129-31. doi: 10.1213/XAA.0000000000000363. PMID 27513972
- [Background] La Colla L, Ben-David B, Merman R. Quadratus Lumborum Block as an Alternative to Lumbar Plexus Block for Hip Surgery: A Report of 2 Cases. A A Case Rep. 2017 Jan 1;8(1):4-6. doi: 10.1213/XAA.0000000000000406. PMID 28036319
- [Background] Adhikary SD, Short AJ, El-Boghdadly K, Abdelmalak MJ, Chin KJ. Transmuscular quadratus lumborum versus lumbar plexus block for total hip arthroplasty: A retrospective propensity score matched cohort study. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):372-378. doi: 10.4103/joacp.JOACP_335_17. PMID 30386022
- [Background] Børglum J, Moriggl B, Jensen K, Lønnqvist P, Christensen AF, Sauter A, Bendtsen TF. Ultrasound-guided transmuscular quadratus lumborum blockade. British Journal of Anaesthesia 111:eLetters Supplement, 2013.
- [Background] Winnie AP, Ramamurthy S, Durrani Z, Radonjic R: Plexus blocks for lower extremity surgery: New answers to old problems. Anesth Review 1974; 1:11
- [Derived] Polania Gutierrez JJ, Ben-David B, Rest C, Grajales MT, Khetarpal SK. Quadratus lumborum block type 3 versus lumbar plexus block in hip replacement surgery: a randomized, prospective, non-inferiority study. Reg Anesth Pain Med. 2021 Feb;46(2):111-117. doi: 10.1136/rapm-2020-101915. Epub 2020 Nov 11. PMID 33177220

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.8) | 68.6 (11.8) | 67.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 12 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 16 | 19 | 35
  African American | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Pain at Rest After Surgery
Description: Visual Analog Scale (VAS) score (0-10, 0 means no pain, 10 means the worst pain) of pain at rest. A higher score means worse outcomes.
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 3.4 (3.0) | 3.6 (1.9)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — The margin of non-inferiority is 0.5. The true difference between the means is assumed to be -0.2. The significance level (alpha) of the test is 0.05. The data are drawn from populations with standard deviations of 0.7 and 0.3 (PASS 15 Power Analysis and Sample Size Software (2017). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass); p = .770, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pain With Movement After Surgery
Description: Visual Analog Scale (VAS) score (0-10, 0 means no pain, 10 means the worst pain) of pain with movement. A higher score means worse outcomes.
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 4.9 (3.2) | 4.7 (2.0)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .826, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Pain at Rest After Surgery
Description: as for outcome 1
Time Frame: 12 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 3.0 (2.9) | 2.8 (2.0)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .859, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Pain With Movement After Surgery
Description: as for outcome 2
Time Frame: 12 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 4.5 (2.8) | 4.6 (2.1)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .904, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Pain at Rest After Surgery
Description: as for outcome 1
Time Frame: 24 hours after surgery
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 2.8 (2.6) | 1.8 (1.5)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .122, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Pain With Movement After Surgery
Description: as for outcome 2
Time Frame: 24 hours after surgery
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 4.9 (2.8) | 4.3 (1.8)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .379, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Pain During Physical Therapy
Description: as for outcome 2
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
score on a scale | 4.3 (2.5) | 4.2 (1.3)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .881, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Total Opioid Consumption During 24 Hours After Surgery
Description: Narcotics will be converted to oral morphine equivalents
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mg oral morphine equivalents
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
mg oral morphine equivalents | 14.0 (9.3) | 14.7 (10.7)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .818, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Postoperative Time to Accomplish Walking 100 Feet
Description: This measurement is from T0 being out of surgery room time to the point at which the participant was able to walk 100 feet during the first day post-surgery. Values were abstracted from the patient medical records.
Time Frame: within 24 hours after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
minutes | 1449.1 (760.7) | 1358.3 (715.5)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .678, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Block Procedure Duration
Description: Duration that the patient underwent the block procedure during surgery in minutes
Time Frame: during surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
minutes | 11.7 (6.1) | 6.6 (4.7)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .002, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Patients With Postoperative Quadriceps Weakness
Description: patients who report having post-surgical quadriceps weakness.
Time Frame: 12 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
Participants | 15 | 6
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .007, Chi-squared

12. Secondary Outcome: Total Acetaminophen Consumption During 24 Hours After Surgery
Description: Patient electronic medical records were reviewed for total acetaminophen consumption during 24 hours after surgery in milligrams (mg)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
milligrams (mg) | 2782.6 (902.3) | 3087.0 (949.3)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .271, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Total Celecoxib Consumption During 24 Hours After Surgery
Description: Patient electronic medical records were reviewed for total celecoxib consumption during 24 hours after surgery in milligrams (mg)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
milligrams (mg) | 191.3 (185.7) | 178.3 (180.8)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .810, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Total Ketorolac Consumption During 24 Hours After Surgery
Description: Patient electronic medical records were reviewed for total ketorolac consumption during 24 hours after surgery in milligrams (mg)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
milligrams (mg) | 9.8 (17.3) | 12.4 (24.2)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .676, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Total Gabapentin Consumption During 24 Hours After Surgery
Description: Patient electronic medical records were reviewed for total gabapentin consumption during 24 hours after surgery in milligrams (mg)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
milligrams (mg) | 382.6 (238.7) | 395.7 (481.9)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .908, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Total Oral Ketamine Consumption During 24 Hours After Surgery
Description: Patient electronic medical records were reviewed for total oral ketamine consumption during 24 hours after surgery in milligrams (mg)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
milligrams (mg) | 7.4 (12.5) | 13.5 (22.9)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .270, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Opioid Consumption During 0-6 Hours After Surgery
Description: Narcotics will be converted to oral morphine equivalents
Time Frame: 6 hours after surgery
Measure: Mean (Standard Deviation); unit: mg oral morphine equivalents
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
mg oral morphine equivalents | 3.4 (3.2) | 6.3 (4.5)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .015, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Opioid Consumption During 6-12 Hours After Surgery
Description: Narcotics will be converted to oral morphine equivalents
Time Frame: 6-12 hours after surgery
Measure: Mean (Standard Deviation); unit: mg oral morphine equivalents
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
mg oral morphine equivalents | 5.0 (4.2) | 3.4 (4.0)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .203, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Opioid Consumption During 12-24 Hours After Surgery
Description: Narcotics will be converted to oral morphine equivalents
Time Frame: 12-24 hours after surgery
Measure: Mean (Standard Deviation); unit: mg oral morphine equivalents
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
Number analyzed (Participants) | 23 | 23
mg oral morphine equivalents | 5.7 (4.6) | 5.0 (5.9)
Statistical Analysis 1: Comparison: Lumbar Plexus Block vs Quadratus Lumborum Type 3 Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .672, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Lumbar Plexus Block | Quadratus Lumborum Type 3 Block
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
The study was conducted at a single-center, potentially confounding external validity. Though the desired statistical power was achieved, our sample was still small. More non-inferiority studies are needed to confirm our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03801265/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03801265/SAP_001.pdf